CLINICAL TRIAL: NCT00607308
Title: A Phase 1, Randomized, Placebo-Controlled, Double Blind, Dose-Escalation, Multicenter Study Of The Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, And Immunogenicity Of A Single Intravenous Dose Of PF-04360365 In Japanese Patients With Mild To Moderate Alzheimer's Disease
Brief Title: A Phase I, Single Dose Study Of PF-04360365 In Japanese Patients With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trials Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9951005
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 0.1 mg/kg (Experimental)
  Interventions: Biological: PF-04360365
- 0.5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365
- 1 mg/kg (Experimental)
  Interventions: Biological: PF-04360365
- 5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 10 mg/kg (Experimental)
  Interventions: Biological: PF-04360365

INTERVENTIONS:
Biological: PF-04360365 — Single dose of 0.1 mg/kg IV on Day 1
  Arms: 0.1 mg/kg
Biological: PF-04360365 — Single dose of 0.5 mg/kg IV on Day 1
  Arms: 0.5 mg/kg
Biological: PF-04360365 — Single dose of 1 mg/kg IV on Day 1
  Arms: 1 mg/kg
Biological: PF-04360365 — Single dose of 5 mg/kg IV on Day 1
  Arms: 5 mg/kg
Drug: Placebo — Single dose of placebo IV on Day 1
  Arms: Placebo
Biological: PF-04360365 — Single dose of 10 mg/kg IV on Day 1
  Arms: 10 mg/kg

SUMMARY:
The purpose of this study is to examine the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of a single dose of PF-04360365 in Japanese subjects with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or females of non-childbearing potential, ages 50-85
* Diagnosis of probable Alzheimer's disease, consistent with criteria from both: (1) National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) 2) Text Revision of The Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR)
* Mini-Mental Status Exam score of 16-26 inclusive
* Rosen-Modified Hachinski Ischemia score < or = 4

Exclusion Criteria:

* Diagnosis or history of other dementia or neurodegenerative disorders
* Diagnosis or history of clinically significant cerebrovascular disease
* Specific findings on magnetic resonance imaging (MRI): cortical infarct, micro hemorrhage, multiple white matter lacunes, extensive white matter abnormalities
* History of autoimmune disorders
* History of allergic or anaphylactic reactions

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To examine the safety and tolerability of a single dose of PF-04360365 in Japanese subjects with mild to moderate AD for one year following dosing. | 1 year

SECONDARY OUTCOMES:
To characterize the pharmacokinetic, pharmacodynamic and immunogenicity profile of PF-04360365 for one year following dosing. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Japan (9):
  - Pfizer Investigational Site, Hirosaki, Aomori
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Fukuyama, Hiroshima
  - Pfizer Investigational Site, Tsukuba, Ibaraki
  - Pfizer Investigational Site, Kanazawa, Kanazawa
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Niigata, Niigata
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Kodaira, Tokyo

REFERENCES:
- [Derived] Miyoshi I, Fujimoto Y, Yamada M, Abe S, Zhao Q, Cronenberger C, Togo K, Ishibashi T, Bednar MM, Kupiec JW, Binneman B. Safety and pharmacokinetics of PF-04360365 following a single-dose intravenous infusion in Japanese subjects with mild-to-moderate Alzheimer's disease: a multicenter, randomized, double-blind, placebo-controlled, dose-escalation study. Int J Clin Pharmacol Ther. 2013 Dec;51(12):911-23. doi: 10.5414/CP201816. PMID 24131736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9951005&StudyName=A%20Phase%20I%2C%20Single%20Dose%20Study%20Of%20PF-04360365%20In%20Japanese%20Patients%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease%20